CLINICAL TRIAL: NCT00216996
Title: Study on the Effect of Glutamine Supplemented Nutrition Support on Protein and Glutamine Metabolism in Severely Burned Patients
Brief Title: Effect of Glutamine Supplemented Nutrition Support on Protein and Glutamine Metabolism in Burns
Status: Withdrawn | Type: Observational
Why Stopped: This study was withdrawn (see NCT00181753).
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ronald G. Tompkins, Chief, Burns Service, Massachusetts General Hospital
Other Study IDs: 1999-P-008464; 5P50GM021700-26 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Burns
Keywords: parenteral nutrition; burn injury; stable isotopes; Glutamate Metabolic Kinetics; Glutamine Metabolic Kinetics
MeSH Terms: conditions — Burns; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Burn patients: Receiving standard TPN with or without glutamine enrichment

SUMMARY:
The Total Parenteral Nutrition (TPN)received as part of your routine burn care has optimal levels of protein and sugar, however the best mixture of amino acids for a patient with burn wounds is not yet known. Amino acids occur naturally in the body and the food we eat. The body combines amino acids to make protein. It uses the proteins to do things such as heal wounds, fight infection, and provide energy. We are studying if the body's use of protein is increased after receiving TPN containing the amino acid called glutamine. We hope to learn the best composition of TPN so that the body can more efficiently repair wounded tissues and recover earlier from an acute burn injury.

DETAILED DESCRIPTION:
Human and animal studies have demonstrated that glutamine catabolism exceeds glutamine synthesis in burn patients, resulting in a glutamine-depleted status, which compromises liver function, including glutathione status, proline and arginine homeostasis and whole body protein balance (1). The purpose of this study is to directly quantify glutamine / glutamate kinetics in relation to glutamine / glutamate disposal and whole body amino acid balance, by using stable isotope tracers [1-13C, 15N]leucine and [15N2]urea.

We hypothesize that the enrichment of amino acid mixtures with glutamine will attenuate overall body nitrogen catabolism and better maintain proline and arginine homeostasis.

The purpose of this study it to 1) investigate the effect of glutamine supplemented total parenteral nutrition (TPN) on whole body metabolic and disposal rate of glutamine, and its rate of de novo synthesis in severely burned patients and 2)explore the impact of glutamine supplementation on whole body protein turnover, studied with L-[1-13C, 15N}-leucine, and on the metabolic homeostasis of urea cycle.

ELIGIBILITY:
Inclusion Criteria:

Burn patients being treated at MGH Burn Unit with one or more of the following criteria: 1) >=5% TBSA; 2) inhalation injury; or 3) resting energy expenditure (REE) of >15% of the predicted Basal Metabolic Rate using the Harris-Benedict equation.

Must be receiving total parenteral nutrition in the course of their treatment.

Exclusion Criteria:

Patients with thyroid disease. Patients who are not hemodynamically stable or show unstable vital signs Patients at the stage of major organ failure, e.g. renal and/or liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
This is a study for measuring the protein kinetics for metabolism of the amino acid glutamine. Kinetics will be derived from measurements on blood and air samples taken as part of the study. | 15 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Tompkins, MD, ScD, Principal Investigator — MGH, Shriners Burn Hospital - Boston
Locations (1):
- Massachusetts General Hospital Burn Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Published data will be shared in our publications and directly with an individual researcher when requested.

REFERENCES:
- [Background] Sheridan RL, Prelack K, Yu YM, Lydon M, Petras L, Young VR, Tompkins RG. Short-term enteral glutamine does not enhance protein accretion in burned children: a stable isotope study. Surgery. 2004 Jun;135(6):671-8. doi: 10.1016/j.surg.2003.11.014. PMID 15179374
- [Background] Young VR, Ajami AM. Glutamine: the emperor or his clothes? J Nutr. 2001 Sep;131(9 Suppl):2449S-59S; discussion 2486S-7S. doi: 10.1093/jn/131.9.2449S. PMID 11533293
- [Background] Yu YM, Wagner DA, Walesreswski JC, Burke JF, Young VR. A kinetic study of leucine metabolism in severely burned patients. Comparison between a conventional and branched-chain amino acid-enriched nutritional therapy. Ann Surg. 1988 Apr;207(4):421-9. doi: 10.1097/00000658-198804000-00009. PMID 3128190